CLINICAL TRIAL: NCT03915275
Title: Clinical Impact of 16S rDNA PCR, a Monocentric Retrospective Study
Brief Title: Clinical Impact of 16S rDNA PCR
Acronym: CI16DP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7407
Record Dates: First submitted 2019-04-11; First posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Bacterial Infections
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective of this study is to evaluate the impact of a positive 16S rDNA PCR in various sites on patient's management.

The secondary objectives of the protocol are:

* to evaluate bacterial identification performance
* to evaluate the effect of previous antibiotic therapy
* to analyze the management of discordant results between 16S PCR and culture identification

ELIGIBILITY:
Inclusion Criteria:

* Patients that had a 16S rDNA PCR positive result in Strasbourg University Hospital laboratory from 2014 to 2018
* Patients consent for this analysis of their past medical history
* Legal guardians consent for the analysis of their children's medical history

Exclusion Criteria:

* Patients who express opposition for this study
* Incomplete clinical record

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: tients that had a 16S rDNA PCR positive result in Strasbourg University Hospital laboratory from 2014 to 2018
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-05-01 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Study of the modification of the care of the patients by the use of the 16S PCR | The period from Junuary 1st, 2014 to Dcember 31, 2018 will be examined

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Maladies Infectieuses et Tropicales, Strasbourg, France